CLINICAL TRIAL: NCT00923858
Title: Asymptomatic Cuff Tears: A Model for Pain Development - Part B
Brief Title: The Natural History of Asymptomatic Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB# 201103230; 5R01AR051026 (NIH)
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff; Ultrasound; Pain; Tear Progression
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control - participants from cycles 1 & 2: no intervention. Control group is composed of participants from Cohort I (recruited during our first grant cycle) and from Cohort II (recruited during our second grant cycle). Continued observation is planned for those controls, partial tears and full tears who enrolled in study at age 65 years or younger and have less than 11 years of follow up.
- Cuff Tear Cohort III: These participants are being recruited from our clinical population and have been scheduled to undergo a standard of care rotator cuff repair and post op therapy. One shoulder has been indicated for rotator cuff repair and the contralateral shoulder is asymptomatic. Both shoulders will be monitored.

SUMMARY:
The purpose of this project is to provide information which can help us understand what happens over time to rotator cuff tears. In this study, the investigators will follow a population of people with rotator cuff tears that do not hurt (asymptomatic) and to establish the probability that an asymptomatic rotator cuff tear, identified in the context of contralateral symptoms, will become symptomatic over time. To determine with ultrasound the probability that a rotator cuff tear will enlarge over time. To determine if symptom progression correlates with enlargement of the rotator cuff tear and/or degenerative changes on radiographs. In order to obtain data, study subjects will be recalled for follow-up at 1 year time points over a 5 year period. The study subjects will have repeat physical exam, ultrasound and radiographic examinations. A control group of normal patients will also be followed for comparison.

DETAILED DESCRIPTION:
The specific aims of our study are:

1. To determine the probability that an asymptomatic rotator cuff tear will become symptomatic over time.
2. To determine which epidemiological factors correlate with symptomatic progression.
3. To determine if symptomatic progression correlates with enlargement of the rotator cuff tear as determined at sonography.
4. To determine the value of routine sonographic scanning of the asymptomatic shoulder.

ELIGIBILITY:
Group 1 (Cohorts I & II) Inclusion Criteria:

* Participants who enrolled at age 65 years or younger will remain in the study.
* Less than 11 annual visits of non-operative surveillance of study shoulder.
* Less than 3 annual visits following a rotator cuff repair of study shoulder.

Group 1 (Cohorts I & II) Exclusion Criteria:

* Workman's Compensation claim involving the shoulders.
* Use of crutch, cane or weight-bearing device on study shoulder.
* Moderate or severe glenohumeral arthritis.
* Inflammatory or other disease process affecting neurological/musculoskeletal systems that may impact weight-bearing activities or normal use of upper body.
* Inability to return for routine study visits.
* Traumatic injury to rotator cuff.
* Rotator Cuff Tear greater than 30mm in width.
* Advanced fatty muscle degeneration.

Patients who are currently enrolled but require a shoulder replacement will not remain in the study. Cohorts I & II will now be considered the control group for comparison to those enrolled in this next recruitment period.

Group 2 (Cohort III) Inclusion Criteria:

* Age 65 years or younger.
* Surgical candidate for primary, double-row repair of a rotator.
* Able to comply with post operative therapy protocol.
* Bilateral partial or full thickness rotator cuff tears: one symptomatic requiring surgery and the contralateral shoulder asymptomatic.

Group 2 (Cohort III) Exclusion Criteria:

* Workman's Compensation claim involving the shoulders.
* Use of crutch, cane or weight-bearing device on study shoulder.
* Moderate or severe glenohumeral arthritis.
* Inflammatory or other disease process affecting neurological/musculoskeletal systems that may impact weight-bearing activities or normal use of upper body.
* Inability to return for routine study visits.
* Traumatic injury to rotator cuff.
* Rotator Cuff Tear greater than 30mm in width.
* Advanced fatty muscle degeneration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from orthopaedic surgeon's clinic.
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2005-07-01 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Standardized Shoulder Ultrasound & Radiographs | Through study completion, an average of 1 per year
  The ultrasound involves measurement of rotator cuff tear (if present) and assessment of muscle degeneration. Radiographs will be used to document any bony changes.

SECONDARY OUTCOMES:
American Shoulder & Elbow Survey (ASES) | Through study completion, an average of 1 per year
  Assessment of patient-rated shoulder pain and function/disability. Questions involve activities of daily living that reflect the use of the shoulder & elbow in different planes of motion. Pain and weakness with various activities are also addressed. (Range 0-100, higher scores indicate better outcomes)
Western Ontario Rotator Cuff (WORC) Index | Through study completion, an average of 1 per year
  Disease-specific quality of life questionnaire, evaluating the change in symptoms and functional ability, specific to rotator cuff tendinopathy. (Range: 0-2100, normalized to 0-100, higher scores indicate worst possible symptoms)
Short Form Health Survey (SF-12) | Through study completion, an average of 1 per year
  General health assessment composed of two scales, Physical Component Summary and Mental Component Summary (Range: 0-100, higher scores indicate better health)

OTHER OUTCOMES:
Physical Examination by the study coordinator (Range of motion) | Through study completion, an average of 1 per year
  Research team member measures shoulder range of motion using a goniometer.
Physical Examination by the study coordinator (Strength) | Through study completion, an average of 1 per year
  Research team member measures shoulder strength measured with a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jay D Keener, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgarten KM, Gerlach D, Galatz LM, Teefey SA, Middleton WD, Ditsios K, Yamaguchi K. Cigarette smoking increases the risk for rotator cuff tears. Clin Orthop Relat Res. 2010 Jun;468(6):1534-41. doi: 10.1007/s11999-009-0781-2. Epub 2009 Mar 13. PMID 19283436
- [Background] Bright AS, Torpey B, Magid D, Codd T, McFarland EG. Reliability of radiographic evaluation for acromial morphology. Skeletal Radiol. 1997 Dec;26(12):718-21. doi: 10.1007/s002560050317. PMID 9453105
- [Background] Codman EA, Akerson IB. THE PATHOLOGY ASSOCIATED WITH RUPTURE OF THE SUPRASPINATUS TENDON. Ann Surg. 1931 Jan;93(1):348-59. doi: 10.1097/00000658-193101000-00043. No abstract available. PMID 17866481
- [Background] COTTON RE, RIDEOUT DF. TEARS OF THE HUMERAL ROTATOR CUFF; A RADIOLOGICAL AND PATHOLOGICAL NECROPSY SURVEY. J Bone Joint Surg Br. 1964 May;46:314-28. No abstract available. PMID 14167640
- [Background] Deutsch A, Altchek DW, Schwartz E, Otis JC, Warren RF. Radiologic measurement of superior displacement of the humeral head in the impingement syndrome. J Shoulder Elbow Surg. 1996 May-Jun;5(3):186-93. doi: 10.1016/s1058-2746(05)80004-7. PMID 8816337
- [Background] Dunn WR, Schackman BR, Walsh C, Lyman S, Jones EC, Warren RF, Marx RG. Variation in orthopaedic surgeons' perceptions about the indications for rotator cuff surgery. J Bone Joint Surg Am. 2005 Sep;87(9):1978-84. doi: 10.2106/JBJS.D.02944. PMID 16140812
- [Background] Galatz LM, Ball CM, Teefey SA, Middleton WD, Yamaguchi K. The outcome and repair integrity of completely arthroscopically repaired large and massive rotator cuff tears. J Bone Joint Surg Am. 2004 Feb;86(2):219-24. doi: 10.2106/00004623-200402000-00002. PMID 14960664
- [Background] Goodman RS. Abnormal findings on magnetic resonance images of asymptomatic shoulders. J Bone Joint Surg Am. 1996 Apr;78(4):633. No abstract available. PMID 8609145
- [Background] Goutallier D, Postel JM, Bernageau J, Lavau L, Voisin MC. Fatty muscle degeneration in cuff ruptures. Pre- and postoperative evaluation by CT scan. Clin Orthop Relat Res. 1994 Jul;(304):78-83. PMID 8020238
- [Background] Harryman DT 2nd, Mack LA, Wang KY, Jackins SE, Richardson ML, Matsen FA 3rd. Repairs of the rotator cuff. Correlation of functional results with integrity of the cuff. J Bone Joint Surg Am. 1991 Aug;73(7):982-9. PMID 1874784
- [Background] Hollister MS, Mack LA, Patten RM, Winter TC 3rd, Matsen FA 3rd, Veith RR. Association of sonographically detected subacromial/subdeltoid bursal effusion and intraarticular fluid with rotator cuff tear. AJR Am J Roentgenol. 1995 Sep;165(3):605-8. doi: 10.2214/ajr.165.3.7645478.
- [Background] Kamath G, Galatz LM, Keener JD, Teefey S, Middleton W, Yamaguchi K. Tendon integrity and functional outcome after arthroscopic repair of high-grade partial-thickness supraspinatus tears. J Bone Joint Surg Am. 2009 May;91(5):1055-62. doi: 10.2106/JBJS.G.00118. PMID 19411453
- [Background] Kowalsky MS, Keener JD. Revision arthroscopic rotator cuff repair: repair integrity and clinical outcome: surgical technique. J Bone Joint Surg Am. 2011 Mar;93 Suppl 1:62-74. doi: 10.2106/JBJS.J.01173. PMID 21411687
- [Background] Keyes EL. Observations on Rupture of the Supraspinatus Tendon: Based Upon a Study of Seventy-Three Cadavers. Ann Surg. 1933 Jun;97(6):849-56. doi: 10.1097/00000658-193306000-00007. No abstract available. PMID 17866987
- [Background] Kim HM, Dahiya N, Teefey SA, Keener JD, Yamaguchi K. Sonography of the teres minor: a study of cadavers. AJR Am J Roentgenol. 2008 Mar;190(3):589-94. doi: 10.2214/AJR.07.2960. PMID 18287426
- [Background] Mall NA, Kim HM, Keener JD, Steger-May K, Teefey SA, Middleton WD, Stobbs G, Yamaguchi K. Symptomatic progression of asymptomatic rotator cuff tears: a prospective study of clinical and sonographic variables. J Bone Joint Surg Am. 2010 Nov 17;92(16):2623-33. doi: 10.2106/JBJS.I.00506. PMID 21084574
- [Background] Tashjian RZ, Hollins AM, Kim HM, Teefey SA, Middleton WD, Steger-May K, Galatz LM, Yamaguchi K. Factors affecting healing rates after arthroscopic double-row rotator cuff repair. Am J Sports Med. 2010 Dec;38(12):2435-42. doi: 10.1177/0363546510382835. Epub 2010 Oct 28. PMID 21030564
- [Background] Keener JD, Wei AS, Kim HM, Paxton ES, Teefey SA, Galatz LM, Yamaguchi K. Revision arthroscopic rotator cuff repair: repair integrity and clinical outcome. J Bone Joint Surg Am. 2010 Mar;92(3):590-8. doi: 10.2106/JBJS.I.00267. PMID 20194317
- [Background] Kitay GS, Iannotti JP, Williams GR, Haygood T, Kneeland BJ, Berlin J. Roentgenographic assessment of acromial morphologic condition in rotator cuff impingement syndrome. J Shoulder Elbow Surg. 1995 Nov-Dec;4(6):441-8. doi: 10.1016/s1058-2746(05)80036-9. PMID 8665289
- [Background] Middleton WD. Ultrasonography of the shoulder. Radiol Clin North Am. 1992 Sep;30(5):927-40. PMID 1518937
- [Background] Middleton WD, Edelstein G, Reinus WR, Melson GL, Murphy WA. Ultrasonography of the rotator cuff: technique and normal anatomy. J Ultrasound Med. 1984 Dec;3(12):549-51. doi: 10.7863/jum.1984.3.12.549. PMID 6392585
- [Background] Middleton WD, Payne WT, Teefey SA, Hildebolt CF, Rubin DA, Yamaguchi K. Sonography and MRI of the shoulder: comparison of patient satisfaction. AJR Am J Roentgenol. 2004 Nov;183(5):1449-52. doi: 10.2214/ajr.183.5.1831449. PMID 15505319
- [Background] Middleton WD, Reinus WR, Totty WG, Melson CL, Murphy WA. Ultrasonographic evaluation of the rotator cuff and biceps tendon. J Bone Joint Surg Am. 1986 Mar;68(3):440-50. PMID 3512571
- [Background] Middleton WD, Reinus WR, Totty WG, Melson GL, Murphy WA. US of the biceps tendon apparatus. Radiology. 1985 Oct;157(1):211-5. doi: 10.1148/radiology.157.1.3898217.
- [Background] Middleton WD, Teefey SA, Yamaguchi K. Sonography of the rotator cuff: analysis of interobserver variability. AJR Am J Roentgenol. 2004 Nov;183(5):1465-8. doi: 10.2214/ajr.183.5.1831465. PMID 15505321
- [Background] Milgrom C, Schaffler M, Gilbert S, van Holsbeeck M. Rotator-cuff changes in asymptomatic adults. The effect of age, hand dominance and gender. J Bone Joint Surg Br. 1995 Mar;77(2):296-8. PMID 7706351
- [Background] Miniaci A, Dowdy PA, Willits KR, Vellet AD. Magnetic resonance imaging evaluation of the rotator cuff tendons in the asymptomatic shoulder. Am J Sports Med. 1995 Mar-Apr;23(2):142-5. doi: 10.1177/036354659502300202. PMID 7778695
- [Background] Norwood LA, Barrack R, Jacobson KE. Clinical presentation of complete tears of the rotator cuff. J Bone Joint Surg Am. 1989 Apr;71(4):499-505. PMID 2703509
- [Background] Paletta GA Jr, Warner JJ, Warren RF, Deutsch A, Altchek DW. Shoulder kinematics with two-plane x-ray evaluation in patients with anterior instability or rotator cuff tearing. J Shoulder Elbow Surg. 1997 Nov-Dec;6(6):516-27. doi: 10.1016/s1058-2746(97)90084-7. PMID 9437601
- [Background] Poppen NK, Walker PS. Normal and abnormal motion of the shoulder. J Bone Joint Surg Am. 1976 Mar;58(2):195-201. PMID 1254624
- [Background] Prickett WD, Teefey SA, Galatz LM, Calfee RP, Middleton WD, Yamaguchi K. Accuracy of ultrasound imaging of the rotator cuff in shoulders that are painful postoperatively. J Bone Joint Surg Am. 2003 Jun;85(6):1084-9. doi: 10.2106/00004623-200306000-00016. PMID 12784007
- [Background] Sher JS, Uribe JW, Posada A, Murphy BJ, Zlatkin MB. Abnormal findings on magnetic resonance images of asymptomatic shoulders. J Bone Joint Surg Am. 1995 Jan;77(1):10-5. doi: 10.2106/00004623-199501000-00002. PMID 7822341
- [Background] Sofka CM, Haddad ZK, Adler RS. Detection of muscle atrophy on routine sonography of the shoulder. J Ultrasound Med. 2004 Aug;23(8):1031-4. doi: 10.7863/jum.2004.23.8.1031. PMID 15284460
- [Background] Strobel K, Hodler J, Meyer DC, Pfirrmann CW, Pirkl C, Zanetti M. Fatty atrophy of supraspinatus and infraspinatus muscles: accuracy of US. Radiology. 2005 Nov;237(2):584-9. doi: 10.1148/radiol.2372041612. Epub 2005 Sep 28. PMID 16192321
- [Background] Teefey SA, Rubin DA, Middleton WD, Hildebolt CF, Leibold RA, Yamaguchi K. Detection and quantification of rotator cuff tears. Comparison of ultrasonographic, magnetic resonance imaging, and arthroscopic findings in seventy-one consecutive cases. J Bone Joint Surg Am. 2004 Apr;86(4):708-16. PMID 15069134
- [Background] Teefey SA. Shoulder sonography: why we do it. J Ultrasound Med. 2012 Sep;31(9):1325-31. doi: 10.7863/jum.2012.31.9.1325. No abstract available. PMID 22922611
- [Background] Teefey SA, Middleton WD, Bauer GS, Hildebolt CF, Yamaguchi K. Sonographic differences in the appearance of acute and chronic full-thickness rotator cuff tears. J Ultrasound Med. 2000 Jun;19(6):377-8; quiz 383. doi: 10.7863/jum.2000.19.6.377. PMID 10841058
- [Background] Teefey SA, Middleton WD, Payne WT, Yamaguchi K. Detection and measurement of rotator cuff tears with sonography: analysis of diagnostic errors. AJR Am J Roentgenol. 2005 Jun;184(6):1768-73. doi: 10.2214/ajr.184.6.01841768. PMID 15908528
- [Background] Tyson LL, Crues JV 3rd. Pathogenesis of rotator cuff disorders. Magnetic resonance imaging characteristics. Magn Reson Imaging Clin N Am. 1993 Sep;1(1):37-46. PMID 7584213
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890
- [Background] Yamaguchi K, Sher JS, Andersen WK, Garretson R, Uribe JW, Hechtman K, Neviaser RJ. Glenohumeral motion in patients with rotator cuff tears: a comparison of asymptomatic and symptomatic shoulders. J Shoulder Elbow Surg. 2000 Jan-Feb;9(1):6-11. doi: 10.1016/s1058-2746(00)90002-8. PMID 10717855
- [Background] Yamaguchi K, Tetro AM, Blam O, Evanoff BA, Teefey SA, Middleton WD. Natural history of asymptomatic rotator cuff tears: a longitudinal analysis of asymptomatic tears detected sonographically. J Shoulder Elbow Surg. 2001 May-Jun;10(3):199-203. doi: 10.1067/mse.2001.113086. PMID 11408898
- [Result] Keener JD, Wei AS, Kim HM, Steger-May K, Yamaguchi K. Proximal humeral migration in shoulders with symptomatic and asymptomatic rotator cuff tears. J Bone Joint Surg Am. 2009 Jun;91(6):1405-13. doi: 10.2106/JBJS.H.00854. PMID 19487518
- [Result] Kim HM, Dahiya N, Teefey SA, Keener JD, Galatz LM, Yamaguchi K. Relationship of tear size and location to fatty degeneration of the rotator cuff. J Bone Joint Surg Am. 2010 Apr;92(4):829-39. doi: 10.2106/JBJS.H.01746. PMID 20360505
- [Result] Hamid N, Omid R, Yamaguchi K, Steger-May K, Stobbs G, Keener JD. Relationship of radiographic acromial characteristics and rotator cuff disease: a prospective investigation of clinical, radiographic, and sonographic findings. J Shoulder Elbow Surg. 2012 Oct;21(10):1289-98. doi: 10.1016/j.jse.2011.09.028. Epub 2012 Jan 3. PMID 22217644
- [Result] Keener JD, Steger-May K, Stobbs G, Yamaguchi K. Asymptomatic rotator cuff tears: patient demographics and baseline shoulder function. J Shoulder Elbow Surg. 2010 Dec;19(8):1191-8. doi: 10.1016/j.jse.2010.07.017. Epub 2010 Oct 27. PMID 21030274
- [Result] Kim HM, Dahiya N, Teefey SA, Middleton WD, Stobbs G, Steger-May K, Yamaguchi K, Keener JD. Location and initiation of degenerative rotator cuff tears: an analysis of three hundred and sixty shoulders. J Bone Joint Surg Am. 2010 May;92(5):1088-96. doi: 10.2106/JBJS.I.00686. PMID 20439653
- [Result] Kim HM, Teefey SA, Zelig A, Galatz LM, Keener JD, Yamaguchi K. Shoulder strength in asymptomatic individuals with intact compared with torn rotator cuffs. J Bone Joint Surg Am. 2009 Feb;91(2):289-96. doi: 10.2106/JBJS.H.00219. PMID 19181972
- [Result] Wall LB, Teefey SA, Middleton WD, Dahiya N, Steger-May K, Kim HM, Wessell D, Yamaguchi K. Diagnostic performance and reliability of ultrasonography for fatty degeneration of the rotator cuff muscles. J Bone Joint Surg Am. 2012 Jun 20;94(12):e83. doi: 10.2106/JBJS.J.01899. PMID 22717835
- [Result] Roztocil K, Oliva I, Prerovsky I, Linhart J. The effect of hydroxyethylrutoside and its combination with acetylsalicylic acid in patients with obliterative atherosclerosis. Cor Vasa. 1989;31(2):128-33. PMID 2663343